CLINICAL TRIAL: NCT02901743
Title: "Efficacy of Nonsurgical Periodontal Therapy in Patients With Chronic Renal Disease and Periodontitis: A Biochemical and Microbiological Assay"
Brief Title: Effect on Teeth and Gum Cleaning in Patients With Gum and Kidney Disease
Acronym: ETGPGK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Responsible Party: Principal Investigator, Dr.Thirumalesh, Post Graduate, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D 139206060
Record Dates: First submitted 2016-08-25; First posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Renal Insufficiency Chronic; Chronic Periodontitis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Chronic Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GroupI (Test) (Active Comparator): 20 patients with renal insufficiency chronic and chronic periodontitis underwent scaling and root planing. Clinical parameters( GI,PD,CAL) were assessed at baseline and after 3 months. 2ml blood was drawn to assess serum creatinine levels and urine analysis was done at baseline and after 3 months for urinary albumin: creatinine ratio.Pooled plaque samples were taken at baseline and after 3 months to assess the microbial activity of Treponema Denticola and Tannerella Forsythia by PCR.
  Interventions: Other: Scaling and Root planing
- Group II- (Control) (Active Comparator): 20 patients with chronic periodontitis who underwent scaling and root planing.Clinical parameters(GI,PD,CAL)were assessed at baseline and after 3 months. 2ml blood was drawn to assess seum creatnine levels and urine analysis was done at baseline and after 3 months for serum urinary Albumin:Creatinine ratio.Pooled plaque samples were taken at baseline and after 3 months to assess the microbial activity of Treponema denticola and Tannerella Forsythia by PCR.
  Interventions: Other: Scaling and Root planing

INTERVENTIONS:
Other: Scaling and Root planing — All the patients were asked to use a preprocedural mouthrinse and scaling and rootplaning was done using ultrasonic scalers.

SUMMARY:
The main aim and objective of this study was to evaluate the effects of Non- surgical periodontal therapy on the subgingival microbiota and biochemical parameters in patients with chronic kidney disease and chronic periodontitis.

DETAILED DESCRIPTION:
The study was designed as a Non randomized prospective, interventional clinical trial. The sample size for the study was 40 individuals aged between 35-75 years, equally divided into two groups.

Group I--- Patients with Chronic kidney disease and chronic periodontitis (Test) Group II--- Patients with Chronic periodontitis only (Controls) At baseline both the groups were analyzed for clinical, microbiological and also biochemical parameters and underwent Non-surgical Periodontal treatment (i.e. scaling and root planning). All parameters were reassessed again after 3 months.

A total of 20 patients attending the outpatient wing of Hyderabad Kidney Centre , Malakpet,Hyderabad who were diagnosed clinically with Chronic Kidney disease and willing to participate in the study were included in the study.

Another 20 patients attending the outpatient wing of Department of periodontics, Panineeya Mahavidyalaya Institute of Dental Sciences & Hospital, Hyderabad, diagnosed with Chronic Periodontitis and willing to participate in the study were taken.

Biochemical parameters considered included -serum creatin & urinary albumin: creatin ratio.

Microbiological assay was done by Polymerase chain reaction test (PCR) i.e., pooled plaque samples were taken from both predialysis as well as chronic periodontitis patients.

ELIGIBILITY:
Inclusion Criteria:

* A total of 20 patients diagnosed with Chronic kidney disease, (having abnormal Glomerular filtration rate(GFR) and serum Creatinine levels.) and chronic periodontitis (with at least 15 teeth remaining, and with the presence of ≥4 sites in 3 different teeth having clinical attachment loss (CAL) of ≥ 4mm and bleeding on probing). (Group I)
* 20 patients diagnosed with chronic periodontitis only. (GroupII)

Exclusion Criteria:

* Patients with HIV infection, pregnancy, lupus erythematosus, rheumatoid arthritis, any systemic disorder, periodontal therapy in the preceding 6 months, or on any course of antibiotic prophylaxis for periodontal procedures were excluded from the study

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Levels of Microbiological and Biochemical Parameters | Change in levels of Microbiological and Biochemical parameters were assessed at baseline and 3 months after scaling and rootplaning
  Microbiological assay was done by PCR test i.e., pooled plaque samples were taken from both predialysis as well as chronic periodontitis patients at baseline and 3 months after scaling and root planing.
  Supragingival plaque was removed carefully with a sterile scaler to prevent the contamination of the samples.Sample was harvested from the same site with a sterile Gracey curet 5-6 with one single vertical stroke on the root surface.
  Biochemical assay was done by Modified Jaffe's reaction to assess the levels of Serum Creatinine and urine samples were taken to assess the Albumin:Creatinine ratio

SECONDARY OUTCOMES:
Clinical parameter -Gingival Index (GI) | Change in the GI was assessed at baseline and 3 months after Scaling and rootplaning
  The Gingival index was assessed using a University of Carolina-15 (UNC-15) Probe.
Clinical Parameters-Probing depth(PD) and Clinical attachment levels (CAL) | Change in Pd was assessed at baseline and 3 months after scaling and rootplaning
  The Pd was assessed using UNC-15 Probe
Clinical Parameter- Clinical attachment levels(CAL) | Change in CAL was assessed at baseline and 3 months after scaling and rootplaning
  The CAL was assessed using UNC-15 Probe

CONTACTS AND LOCATIONS:
Overall Officials: Rekha R Koduganti, MDS, Study Director — Panineeya Institute Of Dental Sciences and Research centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher MA, Taylor GW. A prediction model for chronic kidney disease includes periodontal disease. J Periodontol. 2009 Jan;80(1):16-23. doi: 10.1902/jop.2009.080226. PMID 19228085
- [Background] Graziani F, Cei S, La Ferla F, Vano M, Gabriele M, Tonetti M. Effects of non-surgical periodontal therapy on the glomerular filtration rate of the kidney: an exploratory trial. J Clin Periodontol. 2010 Jul;37(7):638-43. doi: 10.1111/j.1600-051X.2010.01578.x. Epub 2010 May 25. PMID 20500539